CLINICAL TRIAL: NCT05326256
Title: Investigation of Trunk Proprioception and the Efficacy of Different Exercise Training on Trunk Proprioception in Adolescent Idiopathic Scoliosis
Brief Title: Trunk Proprioception in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Merve Karatel, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/008
Record Dates: First submitted 2022-02-24; First posted 2022-04-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
Keywords: scoliosis; adolescent; proprioception; exercise
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in the training groups and the statistical assessor will not be informed about which group the individuals belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSSE Group (Experimental): Physiotherapy Scoliosis Specific Exercises (PSSE), 45-minute exercise session with the supervisor, twice a week for 12 weeks
  Interventions: Other: Exercise training- PSSE
- Vestibular Exercise Group (Experimental): Vestibular exercises to be added to PSSE exercises, 45-minute exercise session with the supervisor, twice a week for 12 weeks
  Interventions: Other: Exercise training- PSSE with vestibular exercises

INTERVENTIONS:
Other: Exercise training- PSSE — Barcelona Scoliosis Physical Therapy School (BSPTS) method exercises
  Arms: PSSE Group
Other: Exercise training- PSSE with vestibular exercises — Vestibular exercises added to Barcelona Scoliosis Physical Therapy School (BSPTS) exercises
  Arms: Vestibular Exercise Group

SUMMARY:
Aims of this clinical research:

* To investigate trunk proprioception in all three planes in individuals with adolescent idiopathic scoliosis (AIS),
* To investigate the pelvis orientation sense in all three planes in individuals with adolescent idiopathic scoliosis,
* To investigate whether trunk proprioception and pelvis orientation sense are improved with Physiotherapy Scoliosis Specific Exercises (PSSE) in AIS,
* To investigate whether trunk proprioception and pelvis orientation sense are improved with vestibular exercise training to be added to PSSE exercises in AIS,
* Comparison of the effects of different exercise training on trunk proprioception and pelvis orientation sense in AIS
* To examine the parameters that may be associated with the improvement of trunk proprioception of different exercise training (health-related quality of life, perception of cosmetic deformity, scoliosis-related clinical features such as Cobb angle, axial trunk rotation, curve type, etc.).

DETAILED DESCRIPTION:
This clinical study includes examining trunk proprioception and pelvis orientation in all three planes, pain, flexibility, health-related quality of life, perception of cosmetic deformity, dynamic balance, and the effectiveness of different exercise training in individuals aged 10-18 years with a diagnosis of adolescent idiopathic scoliosis and who have PSSE indication.

As the control group; healthy peers with the same characteristics as the exercise groups will be included and they have a negative result of Adam's forward bending test, they do not have any postural disorders.

As a result of the randomization to be applied to the individuals, they will be divided into two groups: PSSE exercise group and vestibular exercise group (vestibular exercises added to PSSE exercises).

Initial assessments will be given to all individuals. Exercise training groups will participate in a 45-minute exercise session with the supervisor, twice a week for 12 weeks. Before exercise training, individuals and their parents will be informed about education and daily life activities.

Apart from the exercises performed under the supervision of a physiotherapist, individuals will be given a home exercise program, and the family and the individual will be asked to keep a diary to evaluate their compliance with the exercise, and the exercise compliance will be evaluated with a phone call every week.

When the exercise training is completed, the training groups will be evaluated as post-training assessments.

In the statistical analysis of data; the values of the control group will be used as normative and will be compared with the data of individuals with scoliosis. The data of the training groups before and after the training program will be compared, and the data of the different exercise groups will be compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adolescent idiopathic scoliosis,
* Aged 10-18,
* Have Physiotherapy Scoliosis Specific Exercises (PSSE) indications,
* Individuals and her/his parents volunteered to participate in the study.

Exclusion Criteria:

* Any contraindication that will prevent the individual from participating to exercise training,
* Have had spinal surgery before,
* Have any mental problems,
* The fact that scoliosis is not idiopathic but has arisen for different reasons (neurological, congenital, etc.),
* The apex of the curve is thoracal-6 vertebrae and above,
* Any neurological, psychiatric, muscular, rheumatic, renal, cardiovascular, pulmonary, tumoral, or orthopedic disease.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change of Trunk Proprioception | Baseline, after the 12 weeks of exercise training
  Thoracic position sense is measured by active angle reproduction using GyKo (Microgate, Bolzano, Italy) inertial system. The system component is located on the trunk at the level of C7-T1 vertebrae. The individual to be measured is standing, for example, the individual to flexion the trunk to 30 degrees and is shown to target angle. Then, the individual is asked to close his eyes and come to the target angle actively. The measurement is repeated 3 times. All data are read from the screen.
Change of Pelvis Orientation Sense | Baseline, after the 12 weeks of exercise training
  Pelvis orientation sense is measured by active angle reproduction using GyKo (Microgate, Bolzano, Italy) inertial system. The system component is located on the lumbar area at the level of the S1 vertebrae. The individual to be measured is standing, performs the anterior-posterior pelvic tilt motion in her/his pelvis, and is shown to target angle. Then, the individual is asked to close his eyes and come to the target angle actively. The measurement is repeated 3 times. All data are read from the screen.
Change of Dynamic balance, spatial orientation | Baseline, after the 12 weeks of exercise training
  Assement of dynamic balance with Fukuda-Utenberger stepping test
Change of Cosmetic Deformity Perception | Baseline, after the 12 weeks of exercise training
  Perception of cosmetic deformity assessment with Walter Reed Visual Evaluation Scale and Turkish version of The Spinal Appearance Questionnaire (SAQ)
Change of Cosmetic Deformity Perception according to Individual, Parent and Physiotherapist | Baseline, after the 12 weeks of exercise training
  Perception of cosmetic deformity assessment with Turkish version of The Spinal Appearance Questionnaire (SAQ)
Change of Health-Related Quality of Life | Baseline, after the 12 weeks of exercise training
  Health-Related Quality of Life Assessment with Turkish version of Scoliosis Research Society-22 (SRS-22) Questionnaire
Change of Body Asymmetry | Baseline, after the 12 weeks of exercise training
  Body asymmetry assessment with POTSI (Postural Trunk Symmetry Index)

SECONDARY OUTCOMES:
Enroll of the Cobb Angle | Baseline, after the 12 weeks of exercise training
  The Cobb angle is measured on postero-anterior full spine radiographs as the standard method of quantifying the amount of lateral deviation of the spine.
Enroll of the Risser sign | Baseline, after the 12 weeks of exercise training
  Risser sign is observed that the state of ossification of the iliac apophysis on radiographs as the standard method of quantifying the skeletal maturity.
Enroll of the clinical features of scoliosis | Baseline, after the 12 weeks of exercise training
  The classification of Lenke, SRS (Scoliosis Research Society), and BSPTS (Barcelona Scoliosis Physical Therapy School) are determined according to individual's radiographs, results of Adam's forward bending test, and orientation of the trunk position regarding pelvis.
Change of Angle of Trunk Rotation | Baseline, after the 12 weeks of exercise training
  Angle of trunk rotation is measured with scoliometer on Adam's forward bending test regarding the size of the hump of the trunk.
Change of Pain | Baseline, after the 12 weeks of exercise training
  Pain assessment with Visual Analogue Scale
Change of Flexibility | Baseline, after the 12 weeks of exercise training
  Flexibility assessment with forward and side bending test
Evaluation of exercise training compliance | Once a week for 12 weeks
  The compliance of the home exercise program is followed by weekly phone calls with the individual and their parents. At the end of the research, the amount of exercise compliance of the individuals will be determined according to the calculation of recommended and performing exercises.

OTHER OUTCOMES:
Change of Quality of Life according to brace- The Brace Questionnaire | Baseline, after the 12 weeks of exercise training
  In individuals using brace:Turkish version of the Brace Questionnaire (BrQ) is used. The minimum score is 20 and the maximum score is 100 and also, high scores indicate a better quality of life in this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided